CLINICAL TRIAL: NCT02771574
Title: A Phase 2 Multi-Ascending Dose Trial to Assess the Efficacy, Tolerability and Pharmacokinetic Profile of Exendin (9-39) in Patients With Post-bariatric Hyperinsulinemic Hypoglycemia
Brief Title: Efficacy, Tolerability and Pharmacokinetics of Subcutaneous Exendin (9-39) in Patients With Post Bariatric Hypoglycemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tracey McLaughlin (Other)
Collaborators: Eiger BioPharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Tracey McLaughlin, Associate Professor of Medicine (Endocrinology), Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 36673
Record Dates: First submitted 2016-05-06; First posted 2016-05-13 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Post Bariatric Hypoglycemia
Keywords: Bariatric surgery complications; Glucose Metabolism Disorders; Exendin (9-39); GLP-1
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — exendin (9-39)

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: Lyo avexitide 0.05 mg/kg (Experimental): Participants will receive lyophilized avexitide (Lyo avexitide) twice daily for 3 days
  Interventions: Drug: Lyo avexitide
- Part A: Lyo avexitide 0.15 mg/kg (Experimental): Participants will receive Lyo avexitide twice daily for 3 days
  Interventions: Drug: Lyo avexitide
- Part A: Lyo avexitide 0.35 mg/kg (Experimental): Participants will receive Lyo avexitide twice daily for 3 days
  Interventions: Drug: Lyo avexitide
- Part A: Lyo avexitide 0.46 mg/kg (Experimental): Participants will receive Lyo avexitide twice daily for 3 days
  Interventions: Drug: Lyo avexitide
- Part B: Liq avexitide 0.38 (±0.03) mg/kg (Experimental): Participants will receive liquid avexitide (Liq avexitide) twice daily for 3 days
  Interventions: Drug: Liq avexitide

INTERVENTIONS:
Drug: Lyo avexitide — Lyophilized avexitide (Lyo avexitide) administered subcutaneously (sc)
  Other Names: Exendin (9-39)
  Arms: Part A: Lyo avexitide 0.05 mg/kg; Part A: Lyo avexitide 0.15 mg/kg; Part A: Lyo avexitide 0.35 mg/kg; Part A: Lyo avexitide 0.46 mg/kg
Drug: Liq avexitide — Liquid avexitide (Liq avexitide) administered subcutaneously (sc)
  Other Names: Exendin (9-39)
  Arms: Part B: Liq avexitide 0.38 (±0.03) mg/kg

SUMMARY:
This study is designed to evaluate the efficacy, safety and pharmacokinetics of subcutaneous exendin (9-39) in subjects with post-bariatric hypoglycemia. Development of this subcutaneous formulation of exendin (9-39) would represent a targeted therapeutic approach for this rare disease with unmet clinical need.

DETAILED DESCRIPTION:
Post-Bariatric Hypoglycemia (PBH) is a rare, but increasingly reported disease occurring after bariatric surgery, characterized by severe hypoglycemic episodes accompanied by symptoms of hypoglycemia. At the moment, no medical therapies have been developed for this disorder, but the clinical need is great. The major contributory factor is thought to be an exaggerated secretion of glucagon-like peptide-1 (GLP-1) due to altered nutrient transit after bariatric surgery. GLP-1 is an incretin hormone secreted primarily by the distal ileum that contributes to postprandial glucose regulation. Exendin (9-39) is a specific GLP-1 receptor antagonist, that when given via continuous IV infusion, has been shown to effectively prevent postprandial hypoglycemia and reduce symptoms of hypoglycemia in patients with PBH. This study is designed to assess the efficacy, safety and pharmacokinetic profile of a novel subcutaneous formulation of exendin (9-39).

ELIGIBILITY:
Inclusion Criteria:

* Post-bariatric surgery more than 6 months prior to signing the informed consent
* Reported history of Whipple's triad: the occurrence of hypoglycemic symptoms associated with a capillary blood glucose of ≤55 mg/dL, and resolution with glucose or carbohydrate administration.
* Symptomatic hypoglycemia during the baseline/screening oral glucose tolerance test (OGTT), as defined by the presence of plasma glucose ≤55 mg/dL with concomitant autonomic and/or neuroglycopenic symptoms.

Exclusion Criteria:

* Patients currently using sulfonylureas or other medications that may interfere with glucose metabolism within 5 half-lives of drug.
* Participation in any clinical investigation within 4 weeks prior to dosing
* History of or current insulinoma
* Active infection or significant acute illness within 2 weeks prior to dosing
* Female patients who are pregnant or lactating
* Women of childbearing potential and not utilizing effective contraceptive methods
* Inadequate end organ function

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Tan, MD, Principal Investigator — Clinical Assistant Professor
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tan M, Lamendola C, Luong R, McLaughlin T, Craig C. Safety, efficacy and pharmacokinetics of repeat subcutaneous dosing of avexitide (exendin 9-39) for treatment of post-bariatric hypoglycaemia. Diabetes Obes Metab. 2020 Aug;22(8):1406-1416. doi: 10.1111/dom.14048. Epub 2020 May 4. PMID 32250530

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Lyo Avexitide 0.5 mg/kg: Lyophilized avexitide (Lyo avexitide) administered subcutaneously (sc) twice daily for 3 days
- Part A: Lyo Avexitide 0.15 mg/kg; Part A: Lyo Avexitide 0.35 mg/kg; Part A: Lyo Avexitide 0.46 mg/kg: Lyo avexitide administered sc twice daily for 3 days
- Part B: Liq Avexitide 0.38 (±0.03) mg/kg: Liquid avexitide (Liq avexitide) administered sc twice daily for 3 days
Period: Lyo Avexitide Dose Level 1 (3 Days)
Arm/Group | Part A: Lyo Avexitide 0.5 mg/kg | Part A: Lyo Avexitide 0.15 mg/kg | Part A: Lyo Avexitide 0.35 mg/kg | Part A: Lyo Avexitide 0.46 mg/kg | Part B: Liq Avexitide 0.38 (±0.03) mg/kg
Started | 3 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Lyo Avexitide Dose Level 2 (3 Days)
Arm/Group | Part A: Lyo Avexitide 0.5 mg/kg | Part A: Lyo Avexitide 0.15 mg/kg | Part A: Lyo Avexitide 0.35 mg/kg | Part A: Lyo Avexitide 0.46 mg/kg | Part B: Liq Avexitide 0.38 (±0.03) mg/kg
Started | 0 | 5 | 0 | 0 | 0
Completed | 0 | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Lyo Avexitide Dose Level 3 (3 Days)
Arm/Group | Part A: Lyo Avexitide 0.5 mg/kg | Part A: Lyo Avexitide 0.15 mg/kg | Part A: Lyo Avexitide 0.35 mg/kg | Part A: Lyo Avexitide 0.46 mg/kg | Part B: Liq Avexitide 0.38 (±0.03) mg/kg
Started | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Lyo Avexitide Dose Level 4 (3 Days)
Arm/Group | Part A: Lyo Avexitide 0.5 mg/kg | Part A: Lyo Avexitide 0.15 mg/kg | Part A: Lyo Avexitide 0.35 mg/kg | Part A: Lyo Avexitide 0.46 mg/kg | Part B: Liq Avexitide 0.38 (±0.03) mg/kg
Started | 0 | 0 | 0 | 3 | 0
Completed | 0 | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Liq Avexitide (3 Days)
Arm/Group | Part A: Lyo Avexitide 0.5 mg/kg | Part A: Lyo Avexitide 0.15 mg/kg | Part A: Lyo Avexitide 0.35 mg/kg | Part A: Lyo Avexitide 0.46 mg/kg | Part B: Liq Avexitide 0.38 (±0.03) mg/kg
Started | 0 | 0 | 0 | 0 | 5
Completed | 0 | 0 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A: Lyo Avexitide 0.05 mg/kg; Part A: Lyo Avexitide 0.15 mg/kg; Part A: Lyo Avexitide 0.35 mg/kg; Part A: Lyo Avexitide 0.46 mg/kg: Lyo avexitide administered sc twice daily for 3 days
- Part B: Liq Avexitide 0.38 mg/kg: Liq avexitide administered sc twice daily for 3 days
- Total: Total of all reporting groups
Arm/Group | Part A: Lyo Avexitide 0.05 mg/kg | Part A: Lyo Avexitide 0.15 mg/kg | Part A: Lyo Avexitide 0.35 mg/kg | Part A: Lyo Avexitide 0.46 mg/kg | Part B: Liq Avexitide 0.38 mg/kg | Total
Number analyzed (Participants) | 3 | 5 | 3 | 3 | 5 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 3 | 3 | 5 | 19
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (14.1) | 50.2 (12.7) | 41.3 (14.6) | 44.7 (10.6) | 48.0 (13.8) | 46.7 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 3 | 3 | 5 | 19
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 0 | 3 | 7
  Not Hispanic or Latino | 2 | 4 | 1 | 3 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 5 | 3 | 2 | 5 | 18
  More than one race | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 3 | 3 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Nadir Glucose
Description: Nadir glucose at baseline and at Day 3 of treatment during oral glucose tolerance test (OGTT).
Time Frame: Day 3 (time zero then every 30 minutes until 180 minutes or gylcemic rescue was required)
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Part A: Lyo Avexitide 0.5 mg/kg; Part A: Lyo Avexitide 0.15 mg/kg; Part A: Lyo Avexitide 0.35 mg/kg; Part A: Lyo Avexitide 0.46 mg/kg: Lyo avexitide administered sc twice daily for 3 days
- Part A: Lyo Avexitide 0.35 mg/kg and 0.46 mg/kg Groups: Lyo avexitide administered sc twice daily for 3 days
  This reporting group is a pooled analysis of data from the Part A: Lyo avexitide 0.35 mg/kg and 0.46 mg/kg groups.
- Part B: Liq Avexitide 0.38 (±0.03) mg/kg: Liq avexitide administered sc twice daily for 3 days
Arm/Group | Part A: Lyo Avexitide 0.5 mg/kg | Part A: Lyo Avexitide 0.15 mg/kg | Part A: Lyo Avexitide 0.35 mg/kg | Part A: Lyo Avexitide 0.46 mg/kg | Part A: Lyo Avexitide 0.35 mg/kg and 0.46 mg/kg Groups | Part B: Liq Avexitide 0.38 (±0.03) mg/kg
Number analyzed (Participants) | 3 | 5 | 3 | 3 | 6 | 5
mg/dL
  Baseline | 41 (5) | 43 (7) | 39 (7) | 42 (4) | 41 (5) | 41 (9)
  Day 3 | 45 (6) | 46 (12) | 51 (3) | 59 (14) | 55 (10) | 60 (13)

2. Secondary Outcome: Change in Composite Symptom Score as a Measure of Treatment Effect
Description: Symptoms of hypoglycemia were assessed using the Edinburgh Hypoglycemia Symptom Scale that measures the intensity of 13 commonly experienced hypoglycemic symptoms, each severity graded on a 6-point Likert scale (0 = not present, 5 = severe). Scores are summed for a composite score ranging from 0 to 65, with higher scores corresponding to more severe hypoglycemia symptoms.
Time Frame: Baseline, Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Lyo Avexitide 0.5 mg/kg | Part A: Lyo Avexitide 0.15 mg/kg | Part A: Lyo Avexitide 0.35 mg/kg | Part A: Lyo Avexitide 0.46 mg/kg | Part A: Lyo Avexitide 0.35 mg/kg and 0.46 mg/kg Groups | Part B: Liq Avexitide 0.38 (±0.03) mg/kg
Number analyzed (Participants) | 3 | 5 | 3 | 3 | 6 | 5
score on a scale
  Baseline | 25 (7) | 12 (4) | 22 (13) | 15 (1) | 19 (9) | 17 (12)
  Day 3 | 25 (11) | 12 (9) | 15 (11) | 7 (3) | 11 (8) | 9 (8)

3. Secondary Outcome: Pharmacokinetics of Subcutaneous Avexitide: Plasma Concentration Prior to Dosing (Co)
Description: Pharmacokinetics of subcutaneous avexitide were assessed on Day 3 of twice daily dosing.
Time Frame: Day 3 (Predose)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: Lyo Avexitide 0.05 mg/kg | Part A: Lyo Avexitide 0.15 mg/kg | Part A: Lyo Avexitide 0.35 mg/kg | Part A: Lyo Avexitide 0.46 mg/kg | Part B: Liq Avexitide 0.38 (±0.03) mg/kg
Number analyzed (Participants) | 3 | 5 | 3 | 3 | 5
ng/mL | 11 (7) | 16 (11) | 4 (2) | 71 (62) | 204 (91)

4. Secondary Outcome: Pharmacokinetics of Subcutaneous Avexitide: Maximum Plasma Concentration (Cmax)
Description: Pharmacokinetics of subcutaneous avexitide were assessed on Day 3 of twice daily dosing.
Time Frame: Day 3 (Predose, and 60, 120, 150, 180, 210, 240, 270, 300, 330, 450, 720 minutes post-dose)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: Lyo Avexitide 0.05 mg/kg | Part A: Lyo Avexitide 0.15 mg/kg | Part A: Lyo Avexitide 0.35 mg/kg | Part A: Lyo Avexitide 0.46 mg/kg | Part B: Liq Avexitide 0.38 (±0.03) mg/kg
Number analyzed (Participants) | 3 | 5 | 3 | 3 | 5
ng/mL | 61 (21) | 156 (54) | 228 (57) | 331 (125) | 359 (195)

5. Secondary Outcome: Pharmacokinetics of Subcutaneous Avexitide: Time of Maximum Plasma Concentration (Tmax)
Description: Pharmacokinetics of subcutaneous avexitide were assessed on Day 3 of twice daily dosing.
Time Frame: Day 3 (Predose, and 60, 120, 150, 180, 210, 240, 270, 300, 330, 450, 720 minutes post-dose)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part A: Lyo Avexitide 0.05 mg/kg | Part A: Lyo Avexitide 0.15 mg/kg | Part A: Lyo Avexitide 0.35 mg/kg | Part A: Lyo Avexitide 0.46 mg/kg | Part B: Liq Avexitide 0.38 (±0.03) mg/kg
Number analyzed (Participants) | 3 | 5 | 3 | 3 | 5
minutes | 270 (30) | 252 (16) | 240 (60) | 190 (46) | 396 (183)

6. Secondary Outcome: Pharmacokinetics of Subcutaneous Avexitide: Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: Pharmacokinetics of subcutaneous avexitide were assessed on Day 3 of twice daily dosing.
Time Frame: Day 3 (Predose, and 60, 120, 150, 180, 210, 240, 270, 300, 330, 450, 720 minutes post-dose)
Measure: Mean (Standard Deviation); unit: ng/mL*min
Arm/Group | Part A: Lyo Avexitide 0.05 mg/kg | Part A: Lyo Avexitide 0.15 mg/kg | Part A: Lyo Avexitide 0.35 mg/kg | Part A: Lyo Avexitide 0.46 mg/kg | Part B: Liq Avexitide 0.38 (±0.03) mg/kg
Number analyzed (Participants) | 3 | 5 | 3 | 3 | 5
ng/mL*min | 21151 (9877) | 51765 (2134) | 77849 (23670) | 129427 (31325) | 147417 (57722)

ADVERSE EVENTS:
Time Frame: Three (3) days per treatment period
Arm/Group | Part A: Lyo Avexitide 0.05 mg/kg | Part A: Lyo Avexitide 0.15 mg/kg | Part A: Lyo Avexitide 0.35 mg/kg | Part A: Lyo Avexitide 0.46 mg/kg | Part B: Liq Avexitide 0.38 (±0.03) mg/kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/3 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 1/3 | 0/5 | 2/3 | 2/3 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Lyo Avexitide 0.05 mg/kg (N=3) | Part A: Lyo Avexitide 0.15 mg/kg (N=5) | Part A: Lyo Avexitide 0.35 mg/kg (N=3) | Part A: Lyo Avexitide 0.46 mg/kg (N=3) | Part B: Liq Avexitide 0.38 (±0.03) mg/kg (N=5)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT02771574/SAP_001.pdf
  • Study Protocol (2016-05-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT02771574/Prot_002.pdf